CLINICAL TRIAL: NCT04919018
Title: Characterizing the Upper Airway Manifestations in Primary Ciliary Dyskinesia and Primary Immunodeficiencies
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Washington University School of Medicine (Other); The Hospital for Sick Children (Other); McGill University (Other); Children's Hospital Medical Center, Cincinnati (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-1170; 5U54HL096458-17 (NIH)
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Primary Ciliary Dyskinesia; Kartagener Syndrome; Primary Immune Deficiency
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood draw for biobanking and future analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Ciliary Dyskinesia (PCD): Subjects with a confirmed diagnosis of PCD
- Primary Immune Deficiency (PID): Subjects with a confirmed diagnosis of PID

SUMMARY:
Though common, morbidities related to upper airway disease in primary ciliary dyskinesia (PCD) and primary immunodeficiencies (PID) have not been fully characterized. These conditions can be difficult to distinguish due to their overlapping phenotypes. The sinonasal and middle ear features are often identified as most problematic by patients and their families, and optimal, highly effective treatment regimens have not been established. The main objective of this project is to characterize and compare the upper airway phenotypes in individuals with confirmed diagnosis of PCD and PID, and to collect critical data to inform the design of future clinical trials of treatment of the upper airway diseases. The investigators anticipate that these investigations will discern the clinical, anatomical, and pathophysiological phenotypes of paranasal sinus disease in PCD and PID, identifying disease endpoints and biomarkers that differentiate these two overlapping disorders. Findings from these studies will also enhance our understanding of middle ear disease and associated hearing loss in a cross-sectional cohort of patients with PCD and PID. Ultimately, the long-term goal of our Consortium is to elucidate underlying phenotypes and genotypes of these diseases, potentially leading to novel therapeutics that will improve the lives of affected individuals. Given the COVID pandemic, certain procedures will have the option to be converted to telehealth visits to ensure compliance with local guidelines and participant safety.

DETAILED DESCRIPTION:
Approximately 200 participants with a diagnosis of PCD (n=100) and PID (n=100) who will each participate in a single study visit will be recruited. 30 percent of participants will be under the age of 12 in both the PCD and PID cohorts. The investigators will use a systematic approach to the diagnostic evaluation of patients in order to identify characteristics which may distinguish between PID and PCD and serve as future clinical trial endpoints. This will include collection of relevant medical history, physical examination, sinonasal quality of life questionnaires, olfactory testing, bilateral audiometry and tympanometry, nasal endoscopy, sinus culture, analysis of mucus composition, Sinus CT scan, nasal nitric oxide measurement and a blood draw.

ELIGIBILITY:
Inclusion Criteria:

Overall inclusion criteria for PCD and PID:

* Ages ≥ 5-45 years.
* Informed consent, and assent from minors.

Inclusion Criteria for PCD:

* Clinical features consistent with PCD plus
* At least one diagnostic test consistent with PCD:

  1. Biallelic pathogenic variants in PCD-associated genes identified by genetic panel testing including deletion/duplication analysis.
  2. Ciliary ultrastructural defect by transmission electron microscopy known to be disease causing, including outer dynein arm defects, outer and inner dynein arm defects, or inner dynein arm defects with microtubular disorganization.

Inclusion Criteria for PID:

- A clinical diagnosis of PID known to be associated with an increased risk of infections, as defined by the European Society of Immunodeficiencies (ESID) registry, AND a genetic confirmation with a known or likely pathogenic variant.

OR a diagnosis of a common variable immunodeficiency (CVID) as defined by the ESID registry:

a. At least one of the following:

i. Increased susceptibility to infection

ii. Autoimmune manifestations

iii. Granulomatous disease

iv. Unexplained polyclonal lymphoproliferation

v. Affected family member with antibody deficiency

b. AND marked decrease of IgG and IgA with or without low IgM levels

c. AND at least one of the following:

i. Poor antibody response to vaccines (and/or absent isohemagglutinins)

ii. Low switched memory B cells (<70 percent of age-related normal value)

d. AND secondary causes of hypogammaglobulinemia have been excluded (e.g., infection, protein loss, medication, malignancy)

e. AND diagnosis established after the 4th year of life

f. AND no evidence of profound T cell deficiency

Exclusion Criteria:

* Inability to undergo study procedures
* Reported increased respiratory symptoms within 3 weeks before the scheduled visit
* Congenital craniofacial abnormalities (cleft lip and/or palate, hemifacial microsomia) that may result in otologic or sinus disease
* Congenital hearing loss
* Diagnosis of Trisomy 21, Kabuki syndrome, DiGeorge anomaly or syndrome, 22q11 deletion syndrome, or CHARGE syndrome
* History of intranasal illicit drug use (i.e. cocaine) or intranasal abuse of over the counter or prescription drugs (i.e. oxycodone, acetaminophen, etc.)
* Pregnancy
* Known selective IgA deficiency, specific antibody deficiency (SPAD), selective IgG subclass deficiency, selective IgM deficiency, mannose-binding lectin deficiency, as well as inborn errors of immunity (IEIs) which are not known to be associated with an increased risk of infections (e.g. autoinflammatory syndromes; unclassified disorders of immune dysregulation)
* Medical condition that is known to cause secondary immunodeficiency, including human immunodeficiency virus (HIV) infection, acquired immunodeficiency syndrome (AIDS), and/or active malignancy
* Patients ever having received gene therapy, hematopoietic stem cell transplant, solid organ transplant, or thymus transplant
* Treatment with targeted immune modulators or immune modifiers
* Treatment with chronic systemic steroids

Ages: 5 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subjects with definite primary ciliary dyskinesia and primary immune deficiencies
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Mean Sinonasal Quality of Life SNOT-22 Score in PCD and PID | During a single 6-hour visit
  SNOT-22 is a subject-completed questionnaire that consists of 22 questions. Each item is rated as follows: 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The total score can range from 0-110, 0 being the best and 110 being the worst.
Mean Quality of Life SN-5 Score in PCD and PID | During a single 6-hour visit
  The Sinus and nasal quality of life survey questionnaire (SN-5) is a quality of life assessment completed by a subject/parent consisting of 5 specific symptoms-related questions (answered on a 7-point Likert scale on the frequency of symptoms, 1=none of the time, 7=all of the time), and 1 general overall quality of life question (answered on a visual analog scale from 0 to 10, worst to best).
Mean Score of Burghart Sniffin' Sticks Threshold Test in PCD and PID | During a single 6-hour visit
  Olfactory function will be evaluated through the Burghart Sniffin' Sticks test which is a validated psychophysical testing method. Sniffin' Sticks test is based on pen-like odor dispensing devices that will be presented to participants. In the the threshold test, subjects will identify an odor at varying concentrations (Continuous Variable Range: 1-16, 1 being the lowest score and 16 being the highest score).
Mean Score of Burghart Sniffin' Sticks Discrimination Test in PCD and PID | During a single 6-hour visit
  Olfactory function will be evaluated through the Burghart Sniffin' Sticks test which is a validated psychophysical testing method. Sniffin' Sticks test is based on pen-like odor dispensing devices that will be presented to participants. In the discrimination test, subjects will select which odor smells different from several options (Continuous Variable Range: 0-16, 0 being the lowest score and 16 being the highest score).
Mean Score of Burghart Sniffin' Sticks Identification Test in PCD and PID | During a single 6-hour visit
  Olfactory function will be evaluated through the Burghart Sniffin' Sticks test which is a validated psychophysical testing method. Sniffin' Sticks test is based on pen-like odor dispensing devices that will be presented to participants. In the identification test, subjects ages 12-45 will identify an odor from four choices (Continuous Variable Range: 0-16, 0 being the lowest score and 16 being the highest score).
Mean Score of Burghart Sniffin' Kids Identification Test in PCD and PID | During a single 6-hour visit
  Olfactory function will be evaluated through the Burghart Sniffin' Sticks test which is a validated psychophysical testing method. Sniffin' Sticks test is based on pen-like odor dispensing devices that will be presented to participants. In the identification test, subjects ages 5-11 will identify an odor from four choices (Continuous Variable Range: 0-14, 0 being the lowest score and 14 being the highest score).
Mean Pure Tone Average Air Conduction in PCD and PID | During a single 6-hour visit
  Audiometry completed by the research team to determine pure tone average in decibels (dB) (Continuous Variable Range: 0-110 dB)
Mean Pure Tone Average Bone Conduction in PCD and PID | During a single 6-hour visit
  Audiometry completed by the research team to determine pure tone average in decibels (dB) (Continuous Variable Range: 0-110 dB)
Characterization of Tympanograms in PCD and PID | During a single 6-hour visit
  Research team will conduct tympanometry and assign one of four types (Type A, Type B, Typc C or large volume) to the completed tympanogram

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Davis, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University, Montreal, Quebec